CLINICAL TRIAL: NCT01308268
Title: Community-based Approach for the Management of Soil-transmitted Helminthiasis in General and Strongyloidiasis in Particular in a Highly Endemic Area
Brief Title: Management of Soil-transmitted Helminthiasis and Strongyloidiasis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidad Nacional de Salta (Other)
Collaborators: Fundación Mundo Sano (Unknown); Albert B. Sabin Vaccine Institute (Other)
Responsible Party: Alejandro Krolewiecki, Instituto de Investigaciones en Enfermedades Tropicales-Universidad Nacional de Salta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIET-05
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-02

CONDITIONS: Helminthiasis; Strongyloides Stercoralis Infection
Keywords: STH; Soil-transmitted Helminthiasis; mass drug administration
MeSH Terms: conditions — Helminthiasis | interventions — Ivermectin; Albendazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ivermectin + Albendazole — Ivermectin: 200µg/kg, single dose, PO + Albendazole 200 (children between 12 and 23 months) or 400 mg (>= 2 years old) single dose, PO

SUMMARY:
The general purpose of the project is to analyse soil-transmitted helminthiases (STH) in a highly endemic area in northern Argentina with a multidisciplinary approach. The specific objectives are to evaluate the local epidemiology of STH, validate a new diagnostic serology method for S. stercoralis and evaluate the efficacy and safety of a mass drug administration regimen with albendazole and ivermectin.

ELIGIBILITY:
Inclusion Criteria:

* All persons that are living in the working area at the time of the intervention and wish to participate in the study.

Exclusion Criteria:

1. All persons that live within the study area but do not want to participate in the study.
2. Pregnant women or women who are likely pregnant.
3. Women during the first post-partum week if they are breastfeeding.
4. Children who weigh less than 15 kg.
5. Persons with a history of hypersensitivity or intolerance to ivermectin, albendazole or to the components that make up those drugs.

Min Age: 1 Year | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2010-12; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Evaluation of local epidemiology of soil-transmitted helminthiases and impact of a mass drug treatment anti-helminthic strategy | 15 months
  Evaluate local epidemiology of STH: frequency of species, prevalence and intensity of infections, groups more affected, morbidity.
  Evaluate the efficacy of a single-dose anti-helminthic regimen for community treatments: albendazole 400 mg + ivermectin 200 mcg/kg.

SECONDARY OUTCOMES:
Validate serology methods for diagnosis of S. stercoralis infection | 15 months
  Compare sensibility, specificity and predictive values of serology for S.stercoralis (ELISA-NIE) with traditional coproparasitological methods
Assess the tolerability and safety of the combination of ivermectin and albendazole | 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Krolewiecki, MD, PhD, Principal Investigator — Universidad Nacional de Salta, Instituto de Investigación en Enfermedades Tropicales
Locations (1):
- Instituto de Investigación en Enfermedades Tropicales, Universidad Nacional de Salta, Orán, Salta Province, Argentina